CLINICAL TRIAL: NCT04929561
Title: The Effect of Breastfeeding Support Provided Via Video-conferencing on Postpartum Anxiety, Breastfeeding Self-Efficacy and Neonatal Outcomes: A Randomized Controlled Trial
Brief Title: The Effect of Breastfeeding Support Provided Via Video-conferencing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Deniz Akyıldız, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Breastfeeding Support
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Breastfeeding; Anxiety Disorders; Neonatal Outcomes
MeSH Terms: conditions — Breast Feeding; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-conferencing group (Experimental): The mothers in the video-conferencing group were counseled via video-conferencing a total of six times (three times a week, at equal intervals) during the first 2 weeks after birth. Each interview was approximately 15-20 minutes. In video-conferencing sessions, the breastfeeding position, the mother's grasping the breast, the baby's latch-on, and sucking duration were observed. Mothers' questions were answered and solutions were offered for breastfeeding problems (sore nipple, engorgement, etc.).
  Interventions: Behavioral: Video-conferencing group
- Control group (No Intervention): The mothers in the control group were given usual care before discharge and no intervention was made after discharge.

INTERVENTIONS:
Behavioral: Video-conferencing group — No intervention
  Other Names: Control group
  Arms: Video-conferencing group

SUMMARY:
A randomized control trial was made to examine the effects of breastfeeding support given by the video-conferencing method in the early postpartum period on anxiety, breastfeeding self-efficiency, and newborn outcomes.

ELIGIBILITY:
Inclusion Criteria:

Infants;

* Born between 37 and 42 weeks
* Without severe congenital anomalies

Mothers;

* A single live birth
* Were 18 years of age or over
* At least primary school graduate
* Did not have a disease that prevents breastfeeding
* Had internet access at home or on the phone
* Could speak and understand the Turkish language.

Exclusion Criteria:

* Situations that cause separation of mother and baby
* Hospitalization of the baby in intensive care
* Inability to answer 3 calls in a video call
* They were determined as those who could not be reached during the home visit for the first and second follow

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The mean postpartum maternal anxiety level (mean ± SD) | at 2 weeks and 4 weeks after delivery
  The primary outcome of this study was the mean postpartum maternal anxiety level (mean ± SD) of the mothers at 2 weeks and 4 weeks after delivery. Maternal anxiety level was assessed using the Postpartum Specific Anxiety Scale. The scale comprises 51 items and 4 sub-dimensions. It means that those who score 73 and below on the scale have low postpartum anxiety levels, those who score between 74 and 100 have a medium level, and those who score 101 and above have a high level of anxiety.
The mean breastfeeding self-efficacy level | at 2 weeks and 4 weeks after delivery
  The other main outcome of the study was the mean breastfeeding self-efficacy level (mean ± SD) measured with the Breastfeeding Self-Efficacy Scale Short Form. The scale is likert type and a total score between 14 and 70 is taken from the scale. The higher the score, the higher the breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Neonatal outcomes-Newborn weight (g) | at 2 weeks and 4 weeks after delivery
  Newborn weight (g) was evaluated using the Follow-up Form at 2 weeks and 4 weeks after delivery
Neonatal outcomes-Hypoglycemia of the newborn | at 2 weeks and 4 weeks after delivery
  Hypoglycemia of the newborn was evaluated using the Follow-up Form at 2 weeks and 4 weeks after delivery.
Neonatal outcomes-Need for phototherapy | at 2 weeks and 4 weeks after delivery
  The need for phototherapy was evaluated using the Follow-up Form at 2 weeks and 4 weeks after delivery
Neonatal outcomes-Respiratory morbidity | at 2 weeks and 4 weeks after delivery
  Respiratory morbidity was evaluated using the Follow-up Form at 2 weeks and 4 weeks after delivery
Neonatal outcomes-illness requiring hospitalization | at 2 weeks and 4 weeks after delivery
  Illness requiring hospitalization was evaluated using the Follow-up Form at 2 weeks and 4 weeks after delivery
Neonatal outcomes-Food intake other than breast milk | at 2 weeks and 4 weeks after delivery
  Food intake other than breast milk was evaluated using the Follow-up Form at 2 weeks and 4 weeks after delivery
Neonatal outcomes-Neonatal death | at 2 weeks and 4 weeks after delivery
  Neonatal death was evaluated using the Follow-up Form at 2 weeks and 4 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Betül Bay, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No